CLINICAL TRIAL: NCT07218718
Title: A Pilot Study Examining the Feasibility of Oral Cryotherapy (Popsicles) in Decreasing Dysgeusia in Patients With Prostate Cancer Receiving Single Agent Taxane Therapy
Brief Title: Oral Cryotherapy to Decrease Taste Changes in Prostate Cancer Patients Receiving Taxane Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24904; NCI-2025-07271 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24904 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Cryotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study statistician will generate a password-protected randomization list to ensure blinding. Following completion of baseline questionnaires, the clinical research associate (CRA) will be informed of the group assignment and notify the participant. The study team is blinded to assignment until this point. The CRA will assist with data collection and will not be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (oral cryotherapy) (Experimental): Patients undergo oral cryotherapy over 75 minutes and suck on a popsicle for 5 minutes before, during, and for 10 minutes post-infusion throughout first taxane chemotherapy cycle, up to 21 days, in the absence of unacceptable toxicity.
  Interventions: Procedure: Oral Cryotherapy; Other: Survey Administration
- Arm II (best practice) (Active Comparator): Patients receive usual care and are encouraged not to consume ice or popsicles throughout their first taxane chemotherapy cycle, up to 21 days, in the absence of unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (best practice)
Procedure: Oral Cryotherapy — Undergo oral cryotherapy
  Arms: Arm I (oral cryotherapy)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether cooling the mouth with popsicles (oral cryotherapy) decreases taste changes in prostate cancer patients receiving taxane chemotherapy. Patients receiving chemotherapy can experience a variety of side effects. Changes in the taste of food is a frequent complaint of patients receiving chemotherapy and is underreported as patients may think that it is unavoidable and not manageable. Taxane-based chemotherapy is thought to be associated with the most taste changes of any chemotherapy. Taste buds contain a specific type of cell, called gustatory cells, that are located on the surface of the tongue, the soft palate (back, muscular part of the roof of the mouth), and the upper part of the esophagus. These cells consist of five basic tastes: salty, sweet, sour, bitter, and umami (or savory). Oral cryotherapy involves cooling the mouth with ice chips, popsicles, or other cold drinks for several minutes before, during, and after chemotherapy causing the tiny blood vessels in the protective linings inside the mouth to narrow. It is thought that this narrowing will reduce blood flow to the cooled areas, thereby decreasing the amount of chemotherapy that is delivered to the fragile protective linings inside the mouth that causes the taste changes. This may be an effective way to decrease taste changes in prostate cancer patients receiving taxane chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess whether use of oral cryotherapy (popsicles) can decrease taste alterations (TAs) during receiving taxane chemotherapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo oral cryotherapy over 75 minutes and suck on a popsicle for 5 minutes before, during, and for 10 minutes post-infusion throughout first taxane chemotherapy cycle, up to 21 days, in the absence of unacceptable toxicity.

ARM II: Patients receive usual care and are encouraged not to consume ice or popsicles throughout their first taxane chemotherapy cycle, up to 21 days, in the absence of unacceptable toxicity.

After completion of study intervention, patients are followed up prior to cycle 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing taxane chemotherapy must be English speaking and have an Eastern Cooperative Oncology Group (ECOG) performance score < 2
* Documented written informed consent of the participant
* ONE of the following diagnoses:

  * Prostate cancer
* Age: At least 18 years of age or older
* Undergoing initial single agent taxane chemotherapy
* Chemotherapy naïve
* Willingness to:

  * Suck on popsicles during chemotherapy infusion
  * Complete baseline and follow-up surveys

Exclusion Criteria:

* Patients with pre-existing taste alterations, oral surgery, or malformation that may interfere with the study procedure will be excluded. Patients receiving oxaliplatin will be excluded due to oral sensitivity of cold fluids during oxaliplatin administration
* Receiving oxaliplatin chemotherapy
* Pre-existing taste alterations
* Previous oral surgery
* Oral malformation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-09-17 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Change in Chemotherapy-induced Taste Alteration Scale (CiTAS) score | Baseline (T1) to prior to cycle 2 (T2) (Cycle length = 21 days)
  The change score of the CiTAS (total score) from T1 to T2 will be compared between two arms using two sample t test or Kruskal-Wallis test whichever is appropriate. The statistical comparison will be conducted using intent-to-treat. Will use linear mixed model for repeated-measures design to evaluate the group-difference in the changes of CiTAS total score. Model will include time (T1, T2), group (the experimental, control group), group × time interaction, and covariates if necessary. Will evaluate the success of the randomization by examining between arm differences in demographic and clinical characteristics. Variables on which there are significant group differences will be further tested to determine if they meet the assumptions of covariates (chi square or t-test).
Change in taste strip perception | Baseline to prior to cycle 2 (Cycle length = 21 days)
  Taste strips will be analyzed with descriptive statistics. For the 5 basic tastes, will note the percentage of patients who could taste salty, sour, bitter, sweet, and umami at baseline and prior to cycle 2 and compare results between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine M Brant, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States